CLINICAL TRIAL: NCT04067713
Title: Plasma Analysis for Response Assessment and to DIrect the manaGement of Metastatic Prostate Cancer
Acronym: PARADIGM
Status: Active, not recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Epic Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: UCL/18/0513
Record Dates: First submitted 2019-07-24; First posted 2019-08-26 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PARADIGM-D: Newly diagnosed metastatic prostate cancer patients starting long term therapy with Docetaxel with androgen deprivation therapy (ADT).
- PARADIGM-A: Newly diagnosed metastatic prostate cancer patients starting long term therapy with Androgen Receptor Signalling Inhibitor (ARSI) drugs with androgen deprivation therapy (ADT).
- PARADIGM-E: Newly diagnosed metastatic prostate cancer patients starting long term therapy with Enzalutamide with androgen deprivation therapy (ADT).

SUMMARY:
This research study is looking into plasma tumour deoxyribonucleic acid (ptDNA), a substance that is shed by cancer cells and can be detected in blood samples. Analysing ptDNA may therefore be able to provide more information about the characteristics of prostate cancer.

This study will involve taking additional blood samples during standard treatment. The samples will be analysed in laboratories for levels of Prostate Specific Antigen (PSA); which gives information on the activity of the cancer; ptDNA; circulating tumour cells (ones that are derived from the cancer) (CTCs) and cells that affect immune system.

The PARADIGM study is not, therefore, testing a new drug. Instead, the study is investigating if a new blood test can provide information about which current treatments for prostate cancer will work best for future patients with this disease.

In the future and PARADIGM's ultimate aim is to identify which of the current treatment options will work best for patients. The research may also identify new opportunities for the development of drugs potentially useful in treating prostate cancer.

DETAILED DESCRIPTION:
In the UK, prostate cancer is the most common cancer in men and with about 1 in 8 men diagnosed with prostate cancer in their lifetime. Up to a third of prostate cancer deaths occur when cancer spreads to other parts of the body known as metastatic prostate cancer, which is a major healthcare burden. Currently, physicians use a maximum of six cycles of Docetaxel and continue Androgen Receptor Signalling Inhibitor (ARSI) drugs until disease progression with long term androgen deprivation therapy (ADT).

There is no early test to indicate if treatment is working for patients with metastatic prostate cancer. Currently Prostate Specific Antigen (PSA) is not sensitive enough to guide treatment alone. Studies in colorectal, lung and prostate cancers have started looking at substance called Plasma tumour deoxyribonucleic acid (ptDNA) and correlated presence of ptDNA will early relapse. Therefore, this study will investigate if the detection of ptDNA after initiating treatment is associated a worse clinical outcome. Our ultimate aim, is to identify which of the current treatment options will work best for patients in the future. This research may also identify new targets for the development of new drugs to test in clinical trials in the future.

Assessments will include blood taken before and during treatment and at cancer progression. In selected centres, an optional Whole Body Magnetic Resonance Imaging (WBMRI) will be performed before and during treatment for those patients who are eligible. Patients will be followed up for a maximum of 10 years at the time they register onto the study. We expect recruitment duration to be 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent
2. Aged 18 or over
3. Polymetastatic disease defined as one of the following:

   i. ≥5 bone metastases ii. ≥1 unequivocal visceral metastases
4. Eastern Cooperative Oncology Group (ECOG) Performance status 0 to 2
5. No medical contra-indications to an Androgen receptor signalling inhibitor (ARSI) or docetaxel (with or without prednisolone).
6. Patients should be either of the following:

   i. Planned to start long-term Luteinizing hormone Releasing Hormone (LHRH) suppression, or ii. Have started long-term LHRH antagonist within the last 14 weeks, or iii. Have started LHRH agonist within the last 16 weeks. When antiandrogens (eg bicalutamide) are used in combination with an LHRH agonist to prevent flare, patients have to have started within 18 weeks of starting antiandrogens..
7. Patients should be planned for addition of docetaxel (PARADIGM-D) or ARSI (PARADIGM-A) within 14 weeks after start of LHRH antagonist ( 16 weeks if LHRH agonist is started without anti-androgen) or 18 weeks from start of anti-androgen with a target of 6 cycles or continuation until progression respectively.
8. No concomitant medical conditions likely to reduce life expectancy.
9. Patient agrees to be followed up in the recruiting centre and to having sequential plasma samples collected as per the study protocol.

Exclusion Criteria:

1 Concurrent or planned for (i.e. prior to development of castration resistance), treatment with oestrogen, radiotherapy or surgery to the primary tumour.

(N.B Patients may also be eligible if randomised to any of the following experimental drugs; PARPi, PD-1/PD-L1 , AKTi, PSMA-lutetium, if given in combination with SOC(i.e. ADT + docetaxel or ARSI) treatment in an open-label clinical trial, or to the placebo arm in an open-label clinical trial following discussion and approval of the CI/delegate. Patients can participate in other observational studies).

2. Prior systemic therapy for prostate cancer other than for LHRHa +/- anti-androgen (started within the time limits defined in inclusion criterion 7).

3. Metastatic brain disease or leptomeningeal disease.

4. Any surgery planned prior to Cycle 4 Day 1 (C4 D1)

5. Other current malignancy or malignancy diagnosed or relapsed within the past 5 years (other than non-melanomatous skin cancer, stage 0 melanoma in situ and non-muscle invasive bladder cancer).

6. Patients who consent to the whole-body magnetic resonance imaging (WBMRI) translational sub-study should have no contraindications to MRI as per local guidelines.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed metastatic prostate cancer patients starting long term therapy with either Androgen Receptor Signalling Inhibitor (ARSI) drugs (PARADIGM A) or Docetaxel (PARADIGM D) with androgen deprivation therapy (ADT).
  This is a UK based trial recruiting from approximately 20 sites over 36 months with a maximum follow up for 10 years. Patients will be screened at Multi disciplinary teams, and patient clinic appointments and those who fulfill eligibility criteria will be offered to take part. They will be given the patient information sheet (PIS) to take away and read and discuss with family and friends. They will be given the opportunity to ask questions before they consent. If the patient wishes, consent can happen on the same day as the PIS was given.
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) and Overall Survival (OS) for PARADIGM-A, PARADIGM-D and PARADIGM-E. | Following completion of cycle 3 or 4 of each patient - PARADIGM A & E, cycle length is 28 days. PARADIGM D, cycle length is 21 days. For OS, 10 years after last patient has been registered
  PFS is defined as the interval from start of ARSI or docetaxel to disease failure as determined by at least one or more of these factors:
  1. Symptomatic or asymptomatic new or unequivocal progression of prior distant metastases confirmed by imaging
  2. Symptomatic progression of cancer in the prostate confirmed by imaging
  3. Serum PSA progression in PARADIGM-D
  4. Death from any cause
  OS is defined as time from start of ARSI or docetaxel with ADT to death from any cause.

SECONDARY OUTCOMES:
Prostate Cancer Specific Survival (PCSS) | 10 years after last patient has been registered
  Prostate Cancer Specific Survival (PCSS) defined as time from start of ARSI or docetaxel with ADT to death from prostate cancer

CONTACTS AND LOCATIONS:
Locations (16):
- United Kingdom (16):
  - Aberdeen Royal Infirmary, Aberdeen
  - Royal Bournemouth Hospital, Bournemouth
  - Velindre University NHS Trust, Cardiff
  - Doncaster and Bassetlaw Teaching Hospitals NHS Foundation Trust, Doncaster
  - Medway NHS Foundation Trust, Gillingham
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - The Princess Alexandra Hospital NHS Trust, London
  - Barts Health NHS Trust, Royal London Hospital, London
  - Kingston Hospital NHS Foundation Trust, London
  - Royal Free London NHS Foundation Trust, London
  - Guy's and St Thomas's NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - University College London Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Undecided